CLINICAL TRIAL: NCT01069926
Title: A Phase I, Multi-center, Open-label, Single Dose Study, to Assess the Pharmacokinetics of AZD1656 and Its Metabolite in Type 2 Diabetes Mellitus Patients With or Without Renal Impairment
Brief Title: To Assess the Pharmacokinetics of AZD1656 and Its Metabolite in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1020C00007
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Glucose Lowering
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — AZD1656

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD1656 — Single dose oral tablet

SUMMARY:
To assess the pharmacokinetics of AZD1656, and its metabolite, in type 2 diabetes mellitus patients with varying degrees of renal impairment and to compare the results with those in patients with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of T2DM for at least 1 year, treated with any OAD or insulin
* Calculated MDRD GFR based on S-creatinine at enrollment should fall within any of the 4 categories: mild , moderate, severe normal

Exclusion Criteria:

* Clinically significant progression of current disease or clinically relevant trauma, as judged by the Investigator, within 2 weeks before the first administration of the IP
* Clinically significant neuropathy according to the Investigator. However subjects with diabetic neuropathy which is not clinically significant according to the Investigator may be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change-from-baseline variables will be calculated for the safety variables listed below, as the post-treatment value minus the value at baseline | The baseline values will be as follows:

SECONDARY OUTCOMES:
To evaluate the safety of AZD1656 in T2DM patients with various degrees of renal impairment. To describe the pharmacodynamics of AZD1656 in T2DM patients with various degrees of renal impairment by assessment of 24-hours glucose profile | blood samples will be collected for up to 48 hours postdose and urine samples for up to 12 hours postdose for measurement of plasma and urine concentrations of AZD1656 and its metabolite

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Principal Investigator — University of Tennessee Medical Center
Locations (4):
- United States (4):
  - Research Site, Orlando, Florida
  - Research Site, Overland Park, Kansas
  - Research Site, Minneapolis, Minnesota
  - Research Site, Knoxville, Tennessee